CLINICAL TRIAL: NCT02819765
Title: Fluid Biomarkers With Deep Phenotyping in Patients With ALS
Brief Title: Deep Phenotyping in Patients With ALS
Status: Completed | Type: Observational
Sponsor: Barrow Neurological Institute (Other)
Collaborators: ALS Association (Other)
Responsible Party: Sponsor
Other Study IDs: ALSA-BIO3; PHX16BN016 (Other: Barrow Neurological Institute)
Record Dates: First submitted 2016-06-07; First posted 2016-06-30 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: ALS; Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Serum Cerebrospinal fluid RNA DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to establish a biorepository and phenotyping database to investigate longitudinal changes in ALS subjects. Blood, including DNA and RNA, cerebrospinal fluid (CSF) and electrophysiologic measures will be collected every 6 months over 1 and a half years. The database and specimen repository will be made available to ALS researchers on a merit basis.

DETAILED DESCRIPTION:
Rationale for the Study

The Northeast ALS Consortium (NEALS) biorepository is an existing resource which has provided scientists with a wide range of samples associated with clinical information. It is primarily cross sectional in nature; longitudinal collections have been associated with a limited set of clinical and functional assessments. The investigators goal is to continue to build this repository with the collection protocol proposed here, to associate biofluid collection with specific measures of upper and lower motor neuron function. This project will compliment others to upgrade the NEALS biorepository infrastructure, including updating the computer systems, expanding the number of sample freezers and establishing a repository in the Western United States, and strengthening the standard operating procedures for the repository. The project also supports existing efforts to expand the biorepository by collecting new blood and spinal fluid samples from people with ALS.

Study Design This is a multicenter, non interventional, longitudinal study in patients with ALS. There will be four (4) subject visits in this study: Baseline, month 6, month 12, and month 18. At each visit, subjects will have biofluids collected, and be evaluated with assessment tools that focus on upper and lower motor neuron burden as well as cognitive function.

Study Objectives and Endpoints The primary objective of the study is to obtain deep phenotyping information on patients studied at regular intervals over 18 months, in conjunction with biofluid collection over that same time period.

The secondary objective of the study is to integrate data from this study to other ongoing projects via the NEALS biorepository, and future collections now being planned.

Endpoints for the study are:

* Motor unit number estimation will be performed on upper extremity muscles using the multipoint incremental technique (MIMUNE);
* Vital capacity, measured using slow vital capacity (SVC).
* Lower motor neuron excitability will be assessed with threshold tracking nerve conduction studies (ttNCS) in the least affected intrinsic hand muscle.
* Cognitive abnormalities will be assessed using the ALS Cognitive Behavior Screen (ALS-CBS);
* Upper motor neuron burden will be assessed using transcranial magnetic stimulation (TMS), employing a paired pulse protocol and recording from the least affected upper extremity intrinsic hand muscle;
* Hand held dynamometry (HHD) will be performed on 10 muscle groups tested bilaterally;
* Global function (ALSFRS-R); and
* Vital capacity, measured using slow vital capacity (SVC).

At each visit, blood will be collected and banked for biomarker discovery; CSF will be collected at baseline, month 6, and at month 18.

Other exploratory objectives of the study (to be performed at Barrow Neurological Institute only) will investigate to the composition of the "pellet" of processed CSF and a novel imaging marker called MRI cytography.

Study Locations Approximately 10 Northeast ALS Consortium (NEALS) Centers in the US will participate in the study. Sites that cannot perform the ttNCS and/or the TMS can still participate.

Number of Planned Subjects Fifty (50) subjects will be in the study. It is estimated that 5 subjects shall be enrolled per site.

Study Population This study will be conducted in subjects who meet the El Escorial criteria of possible, laboratory- supported probable, probable, or definite ALS. Time from diagnosis to study entry must be 24 months or less. At screening, eligible subjects must be at least 18 years old and must provide written informed consent. Detailed criteria will be described in the full protocol.

Duration of Study Active assessment period will be 18 months; a 1-year enrolment period is expected.

ELIGIBILITY:
Inclusion Criteria:

* Participants with sporadic ALS diagnosed as possible, laboratory-supported probable, probable or definite according to the World Federation of Neurology El Escorial criteria.
* Expected to survive >1 year (12 months) after enrollment.
* Male or female, aged 18-75.
* Ability to medically undergo lumbar puncture (LP) as determined by the investigator (i.e., no bleeding disorder, allergy to local anesthetics, prior lumbar surgery which might make LP difficult, a skin infection at or near the LP site, or evidence of high intracranial pressure).
* Willingness and medical ability to comply with scheduled visits, LP for CSF collection, laboratory tests, and other study procedures.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Geographic accessibility to the study site.

Exclusion Criteria:

* Any contraindications to having an LP, including but not limited to: Platelet count <100,000/µL.
* History of bleeding disorder.
* History of intolerance to the LP procedure.
* Evidence of topical or other skin infection at the LP site.
* History of allergy or other adverse reaction to local anesthetics used in the study.
* History of traumatic central nervous system injury or stroke.
* Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment.

Additional criteria for sites performing TMS:

* Inability to perform either TMS or NCS studies due to insufficient motor evoked potential (MEP) or compound muscle action potential (CMAP) amplitude.
* Contraindication to TMS studies including ferromagnetic metal in the head or neck (potentially found in aneurysm clips, implanted medication pumps, implanted brain stimulators, pacemakers, cochlear implants), or history of epilepsy. Dental fillings are permitted.

Additional criteria for sites performing MRI cytography:

* Subjects who have a history of claustrophobia that cannot be adequately controlled.
* Subjects who have a physical limitation related to fitting in the bore of the magnet.
* Subjects who have a history of allergic reaction to contrast agents.
* Subjects with a pacemaker, epicardia pacemaker wires, MRI-incompatible cardiac valve prostheses, MRI-incompatible vascular clips.
* Subjects with MRI-incompatible cochlear implants.
* Subjects with spinal nerve simulators.
* Subjects with an infusion pump.
* Subjects with metallic fragments in the eyes/orbits or in the vicinity of the brain or major neurovascular structures of the body, subjects with an employment history which involves exposure to welding, or subjects who have shrapnel any place in their body.
* Subjects with acute kidney injury or renal insufficiency (eGFR of <20 ml/min/1.73 m^2) as they are at increased risk of Nephrogenic Systemic Fibrosis following administration of gadolinium-based MRI contrast agents.
* Subjects unable to lay supine in the magnet because of orthopnea.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS patient volunteers will be invited to participate in this study by their neurologists either in clinic or at a regular scheduled appointment visit.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
ALS Functional Rating Scale Revised (ALSFRS-R) | Every 6 months through month 18
  The ALSFRS-R is a quickly administered (5 minutes) instrument used to determine subjects' assessment of their capability and independence in 12 functional activities, each rated on an ordinal scale (ratings 0-4).
Slow vital capacity (SVC) | Every 6 months through month 18
  Vital capacity will be measured as slow vital capacity (SVC) using standard technique
Hand held dynamometry (HHD) | Every 6 months through month 18
  Hand held dynamometry (HHD) will be used as a quantitative measure of muscle strength for this study. 10 muscle groups will be examined bilaterally in both upper and lower extremities. Mean and standard deviation for each muscle group will be established from the initial values for each subject in this trial, so that strength determinations can be converted to Z scores and averaged to provide an HHD megascore for both upper and lower extremities.
ALS cognitive behavioral screen (ALS-CBS) | Every 6 months through month 18
  The ALS Cognitive Behavioral Screen (ALS-CBS™) is a short measure of cognition and behavior in patients with Amyotrophic Lateral Sclerosis (ALS). The cognitive section includes commonly used elements of standard testing batteries, consisting of 8 tasks, with a possible total score of 20. It can be administered by a physician or other clinical care staff and takes approximately 5 minutes to complete. The behavioral section (ALS Caregiver Behavioral Questionnaire) is composed of questions sensitive to organic brain changes. It consists of a set of questions that compare changes in personality and behavior since the onset of ALS, as well as yes/no questions about mood, pseudobulbar affect, and fatigue. It is completed by a caregiver, family member or other informant during the same time that the patient completes the cognitive portion. The questionnaire typically takes about 2 minutes to complete.
Multipoint incremental motor unit number estimates (MIMUNE) | Every 6 months through month 18
  MIMUNE is a validated technique to estimate the number of motor units in specific muscles of patients. In this study it will be performed on one intrinsic hand muscle unilaterally throughout the study.
Paired Pulse Stimulation Using Transcranial Magnetic Stimulation (TMS) | Every 6 months through month 18
  TMS is a technique that uses a focused magnetic field to depolarize neurons of interest. By depolarizing motor neurons and measuring the evoked response, an assessment of the neuronal excitability can be determined.
Threshold tracking nerve conduction studies (ttNCS) | Every 6 months through month 18
  ttNCS is a technique that uses stimulation of peripheral motor nerves to measure a variety of variables to determine the excitability of the peripheral motor neurons.

OTHER OUTCOMES:
MRI Cytography | At baseline and at 6 months
  The MRI scan is a non-invasive procedure that uses a powerful magnetic field and radio waves to obtain images of internal organs and tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Shafeeq Ladha, MD, Principal Investigator — Barrow Neurological Institute
Locations (7):
- United States (7):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Spectrum Health, Grand Rapids, Michigan
  - Hospital for Special Surgery (HSS), New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Department of Neurosurgery & Neurology | Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
The data will be part of the Northeast ALS consortium biorepository database.